CLINICAL TRIAL: NCT05087446
Title: Effect of Early Assessment Team for Clarification and Follow-up of Patients Referred to Outpatient Mental Health Care: A Randomized Controlled Trial
Brief Title: Effect of Early Assessment Team for Patients Referred to Outpatient Mental Health Care
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 244508
Record Dates: First submitted 2021-09-13; First posted 2021-10-21 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Mental Disorder
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early assessment group (Experimental)
  Interventions: Behavioral: Early assessment team
- Usual admission procedure group (Active Comparator)
  Interventions: Behavioral: Admission to General psychiatric outpatient clinic

INTERVENTIONS:
Behavioral: Early assessment team — Early assessment team (EAT):The patients receive their first assessment by an early clarification team within a few weeks after the team receiving the referral. The team then decides whether further assessment and/or treatment should be given in the general outpatient clinic, and/or whether any other follow-up may be appropriate. In the first meeting the patient preferably meets two therapists, who conduct a semi-structured interview with focus on health and level of functioning. If considered appropriate, the team may offer a short-term intervention.
  Arms: Early assessment group
Behavioral: Admission to General psychiatric outpatient clinic — Ordinary procedures for admission to an outpatient clinic are followed in accordance with the Norwegian Directorate of Health's national prioritization guide. Referrals are assessed on the basis of severity and placed on a regular waiting list (usually a waiting period of 1-3 months). The patients receive their first personal assessment from a therapist in a general outpatient clinic who takes a position on what is to be initiated and, if necessary, offers further assessment / treatment in accordance with procedures in the outpatient clinics. This is not standardized beyond current practice.
  Arms: Usual admission procedure group

SUMMARY:
Loss of function and incapacity for work as a result of mental disorders are increasing, especially among young people (under 30 years of age), even though the prevalence of mental illness is fairly stable. Many of the patients referred to outpatient mental health care have complex difficulties with both mental and somatic ailments, in addition to difficulties with social conditions related to, for example, education, work, finances and social support. Functional difficulties can come as a result of mental illness. However, it can also be the opposite way; not functioning at work, study or daily life in general can cause mental symptoms and ailments. Many of these people are referred to mental health care even if the basic problem cannot be solved by psychotherapy or medication. Some of the referred patients do not have a psychiatric illness, but a reaction to a stressful and demanding situation and strains over time. Compound health challenges require individualized assessments and clarifications in order to offer the right measures. Traditionally in mental health care, the patient is placed on a waiting list to receive assessment and therapy for a specific condition.

With this background, the investigators believe it is important to early identify the referred patients who will benefit from measures other than traditional assessment and treatment in mental health care. Knowledge of other aid agencies is important to find the right measures at the right time. This is important for the individual patients, who are often young people going to "get started in life". It is also important for the health services because the capacity to provide a good health service is a limited resource. From a societal perspective it is important that the health care offered contributes to reducing social security dependence.

The purpose of this randomized, controlled trial is to compare the effect of traditional management of newly referred patients in outpatient clinics with assessment through an Early Assessment Team. The investigators believe that early assessment may have a positive effect on mental health, quality of life and function. The outcome goals can be summarized as less use of resources in outpatient clinics and society and better function and life for patients.

ELIGIBILITY:
Inclusion Criteria:

* all patients referred to a general psychiatric outpatient clinic
* necessary capacity to consent
* master Norwegian language to such an extent that the patient can understand the written consent

Exclusion Criteria:

* patients that an admission team at the outpatient clinic consider obviously must have a TAU for some time
* patients too healthy to receive specialized mental health care
* patients in need of acute psychiatric assessment
* relevant participants who do not respond digitally or who do not confirm consent in writing within given deadlines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 588 (Estimated)
Dates: Start 2021-10-26 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Work and Social Adjustment Scale (WSAS) | 1 year
  WSAS is a self-report questionnaire with five items covering the following dimensions; influence on work, home management, social leisure activity, private leisure activities and relationships with others. The items are scored from 0 to 8, with a total score from minimum 0 to maximum 40, with lower scores indicating better adjustment.

SECONDARY OUTCOMES:
World Health Organization Well Being Index (WHO-5) | 2, 4, 8, 12, 24 months after enrollment
  The World Health Organization Well Being Index is one of the most widely used measures of subjective psychological well-being that is also a measure of depression. The scale consists of 5 questions about participants well-being experienced during the past 2 weeks. Items are rated on a 6-point scale from 0 (never) to 5 (all the time).
EuroQoL EQ-5D-5L | 2, 4, 8, 12, 24 months after enrollment
  EuroQoL EQ-5D-5L is used to measure health outcomes and perform health economic analyzes. The form consists of 5 questions covering walking, personal care, daily tasks, pain / discomfort and anxiety / depression. In addition, the patient must indicate their own state of health on a VAS scale from 0-100.
Client Satisfaction Questionnaire (CSQ-8) | Through study completion, an average of 1 year
  The measure yields a continuous score on a single factor of general satisfaction. This is derived from eight questions about the quality of service, the kind of service, patients' outcomes and overall satisfaction. The scale is rated on a 4-point response scale.
Clinical Outcome in Routine Evaluation Outcome Measure (CORE-OM) | 12, 24 months after enrollment
  A self-administered questionnaire with 34 items related to the preceding week mapping 4 main areas; well-being (4 elements), problems (12 elements), function (12 elements) og risk (6 elements). All items are scored from "Never" (=0) to "Almost all the time" (=4).
Clinical Outcome in Routine Evaluation Outcome Measure (CORE-10) | 2, 4, 8 months after enrollment
  A self-administered short form of CORE-OM (see outcome 5) with 10 items
The Questionaire about the Process of Recovery (QPR-15) | 2, 4, 8, 12, 24 months after enrollment
  The scale is used to capture peoples' accounts of recovery from severe mental illness. The 15-item version has been recommended for use both in routine clinical work and in research, and it is scored on a 5-point scale from 0 = disagree strongly to 4 = agree strongly).
Occupational status - data extracted from The Norwegian Labour and Welfare Administration (NAV) | 12 and 24 months
  The Norwegian Labour and Welfare Administration (NAV) have data on all citizens working status and sick leaves lasting for more than two weeks. Extracted data will include information such as sick- and disability leaves until 12 and 24 months after enrolment.
Work and Social Adjustment Scale (WSAS) | 2, 4, 8, 24 months after enrollment
  WSAS is a self-report questionnaire with five items covering the following dimensions; influence on work, home management, social leisure activity, private leisure activities and relationships with others. The items are scored from 0 to 8, with a total score from minimum 0 to maximum 40, with lower scores indicating better adjustment.

CONTACTS AND LOCATIONS:
Overall Officials: Jon Helle, MD, Study Chair — Nidelv DPS, Tiller, St.Olavs hospital
Locations (1):
- Nidelv DPS, Tiller, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kvestad CA, Holte IR, Reitan SK, Chiappa CS, Helle GK, Skjervold AE, Rosenlund AMA, Watne O, Brattland H, Helle J, Follestad T, Hara KW, Holgersen KH. Measuring the Effect of the Early assessment Team (MEET) for patients referred to outpatient mental health care: a study protocol for a randomised controlled trial. Trials. 2024 Mar 11;25(1):179. doi: 10.1186/s13063-024-08028-6. PMID 38468321